CLINICAL TRIAL: NCT07041606
Title: Multicenter, Observational, Prospective Study of Molecular Profiling in Advanced and Aggressive Endometrial Cancer Patients and 1-st Line Treatment Approaches in Russian Federation
Brief Title: An Observational Study of Molecular profIling of Advanced and aggRessive ENdometrial Cancer and 1-st Line Treatment Approaches in Russian Federation
Acronym: IREN
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00117
Record Dates: First submitted 2025-06-06; First posted 2025-06-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Multicenter, observational, prospective study of molecular profiling in advanced and aggressive endometrial cancer patients and 1-st line treatment approaches in Russian Federation

DETAILED DESCRIPTION:
This study is national, multi-center, prospective, cohort study to collect real world data of endometrial cancer patients with aggressive advanced (stage III-IV) disease, prevalence of POLEm, dMMR/pMMR, p53abn, HER2, PD-L1, demographic and clinical characteristics and 1-st line (postoperative) treatment approaches in Russian Federation. The study will sequentially include only those patients who have signed the informed consent form (ICF). No additional procedures besides those already used in the routine clinical practice will be applied to the patients.

Study population will consist of patients with newly diagnosed aggressive subtypes of advanced (III-IV stages) EC, with available medical history, biopsy or post-operative archival FFPE tumor samples (blocks). It is estimated that approximately 500 patients will be enrolled in about 30 sites.

In the study there will be two visits carried out according to routine clinical practice. At baseline visit (visit 1) demographic and clinical characteristics and treatment approaches from the date of newly diagnosed advanced (III-IV stages) EC of aggressive subtype will be collected based on the patient's medical records. In case of absence of data required to be collected by the protocol, additional data may be obtained during patient's interview directly and recorded in the source documents related to the visit. For POLEm, dMMR/pMMR, p53abn, HER2, PD-L1 testing, biopsy or post-operative archival FFPE tumor sample (block), will be used. Testing will be performed using immunohistochemistry (IHC) (for MMR, p53, HER2, PD-L1) and next-generation sequencing (NGS) or polymerase chain reaction (PCR) (for POLEm) in central laboratories.

Visit 2 (final visit) will be conducted in 6 months after baseline (±6 weeks) or at progression of the disease (whichever comes first) to collect follow-up data on treatment approaches, and progression (if applicable).

All study data will be entered into electronic case report form (eCRF). The study physician will be responsible for ensuring that all required data is collected and entered into the eCRF.

Overall expected duration of the study (from the first patient inclusion to the final database lock) is about 27 months, or until 500 eligible patients are included to the study and data on these patients are collected (including follow-up data), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥ 18 years old;
2. Signed ICF, including consent for archival FFPE tumor tissue block testing;
3. Newly diagnosed, histologically confirmed, advanced (III-IV stage) EC, with the date of diagnosis of histologically confirmed disease within 4 months before inclusion;
4. Endometrioid type G3 or any non-endometrioid histological type of EC (such as serous carcinoma, clear cell carcinoma, mixed carcinoma, undifferentiated and dedifferentiated carcinoma, carcinosarcoma, others);
5. The presence of biopsy or postoperative archival FFPE tumor sample (block);
6. Availability of source medical documentation.

Exclusion Criteria:

1. Patients participating in clinical (interventional) studies since the diagnosis of histologically confirmed, advanced EC.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients aged ≥ 18 years old;
Study Population: Study population will consist of patients with newly diagnosed aggressive subtypes of advanced (III-IV stages) EC, with available medical history, biopsy or post-operative archival FFPE tumor samples (blocks). It is estimated that approximately 500 patients will be enrolled in about 30 sites.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The rate of POLEm positive status | 24 months
  The rate of Mutation in the exonuclease domain of the Deoxyribonucleic Acid polymerase epsilon (POLE) gene positive status (i.e. detection of pathological variant(s) by Next-Generation Sequencing /Polymerase Chain Reaction), overall and by each variant;
The rate of dMMR status and pMMR status detected by IHC and by combined approach of molecular classification | 24 months
  The rate of Mismatch Repair Deficiency status and Mismatch Repair Proficiency status detected by Immunohistochemistry and by combined approach of molecular classification;
The rate of p53abn positive status detected by IHC and by combined approach of molecular classification | 24 months
  The rate of Abnormal expression of p53 protein positive status detected by Immunohistochemistry and by combined approach of molecular classification;
The rate of PD-L1 positive status detected by IHC | 24 months
  The rate of Programmed Cell Death Ligand 1 positive status (Tumor Area Positivity ≥1%) detected by Immunohistochemistry;
The rate of HER2 expression 3+ detected by IHC | 24 months
  The rate of HER2 expression 3+ detected by Immunohistochemistry according to American Society of Clinical Oncology College of American Pathologists (ASCO CAP) gastric cancer and ASCO CAP guidelines for HER2 testing in Endometrial cancer, and proportion of patients with each result of Immunohistochemistry score (0, 1+, 2+, 3+) on each of the two criteria of evaluation and relationship between them.

SECONDARY OUTCOMES:
Proportion of patients received any 1st line systemic (postoperative) chemotherapy | 33 months
  Proportion of patients received any 1st line systemic (postoperative) chemotherapy, overall and by each regimen/drug;
Duration of the 1st line systemic chemotherapy | 33 months
  Duration of the 1st line systemic (postoperative) chemotherapy (months), No. of cycles of chemotherapy;
Proportion of patients with progression | 33 months
  Proportion of patients with progression according to RECIST 1.1 criteria;
Median time from advanced EC diagnosis to progression | 33 months
  Median time from advanced EC diagnosis to progression (calculated between the date of histologically confirmed advanced EC diagnosis and the date of EC progression according to RECIST 1.1 criteria);
Age at the histologically confirmed diagnosis of aggressive advanced EC | 24 months
  Age at the histologically confirmed diagnosis of aggressive advanced Endometrial cancer
Proportion of patients of different races and ethnicities | 24 months
  Proportion of patients of different races and ethnicities
Proportion of patients with presence of a family oncology history | 24 months
  Proportion of patients with presence of a family oncology history (in first-degree relatives) overall and by each disease;
Proportion of patients with a personal oncology history | 24 months
  Proportion of patients with a personal oncology history overall and by each disease;
Proportion of patients with presence of EC development risk factors | 24 months
  Proportion of patients with presence of EC development risk factors:
  * Obesity (physician-diagnosed or based on BMI>30 kg/m2), current of in the past
  * Smoking status
  * Early menarche (before 12 years)
  * Late menopause (after 55 years)
  * Endometrial hyperplasia
  * Nulliparity
Proportion of patients with each category by ECOG assessment | 24 months
  Proportion of patients with each category by Eastern Cooperative Oncology Group assessment at the inclusion, grades from 0 (Fully active, able to carry on all pre-disease performance without restriction) to 5 (Dead)
Proportion of patients with concomitant diseases | 24 months
  Proportion of patients with concomitant diseases overall and by each disease;
Proportion of patients receiving concomitant therapies | 24 months
  Proportion of patients receiving concomitant therapies overall and by each medicine (by ATC);
Proportion of patients with each clinical stage | 24 months
  Proportion of patients with each clinical stage by TNM (a standard method for classifying the extent of malignant tumors) classification. The size and extent of the primary tumor (T), whether the cancer has spread to nearby lymph nodes (N), and whether the cancer has metastasized to distant parts of the body (M).
Proportion of patients with each clinical stage by FIGO classification | 24 months
  Proportion of patients with each clinical stage by FIGO (The International Federation of Gynecology and Obstetrics (Fédération Internationale de Gynécologie et d'Obstétrique)) classification. FIGO stages are from I (Tumor confined to the corpus uteri) to IVB (Distant metastases, including intra-abdominal metastases and/or inguinal lymph nodes)
Proportion of patients with each histological type of tumour | 24 months
  Proportion of patients with each histological type of tumour
Proportion of patients with each category by grade of differentiation | 24 months
  Proportion of patients with each category by grade of tumor differentiation from G1 (high grade) - highly differentiated) to G3 (low grade) - poorly differentiated;
The rate of each diagnostic methods used in a routine practice in the diagnostics process of EC | 24 months
  The rate of each diagnostic methods used in a routine practice in the diagnostics process of Endometrial cancer

OTHER OUTCOMES:
Proportion of patients underwent surgery | 33 months
  Proportion of patients underwent surgery overall and by each type (if applicable);
Proportion of patients received any radiation therapy | 33 months
  Proportion of patients received any radiation therapy (RT) overall and by each type (if applicable);
Proportion of patients with each radiation area | 33 months
  Proportion of patients with each radiation area (if applicable) (to be calculated in patients who received any RT);
Total RT dose (Gy) by each radiation area | 33 months
  Total radiation therapy (RT) dose (Gray) by each radiation area (to be calculated in patients who received any RT).
Proportion of patients with several biomarkers present at the same time | 24 months
  Proportion of patients with several biomarkers present at the same time, for example, two, three, four, etc. including positive status for POLEm / dMMR/pMMR / p53abn / PD-L1 and positive HER2 expression.

CONTACTS AND LOCATIONS:
Locations (19):
- Russia (19):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Severodvinsk
  - Research Site, Sochi
  - Research Site, Tomsk
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Vladivostok
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org.